CLINICAL TRIAL: NCT02817399
Title: The Effect of Functional Electrical Stimulation on Gait Quality After Anterior Cruciate Ligament Reconstruction
Brief Title: The Effect of Functional Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Collaborators: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16022015
Record Dates: First submitted 2016-03-15; First posted 2016-06-29 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2018-01

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: anterior cruciate ligament reconstruction; Functional Electrical stimulation; Gait analysis; Physical therapy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuro-muscular electrical stimulation (Active Comparator): Active exercises & Neuro-muscular electrical stimulation in a stationary position (lying and/or sitting).
  Interventions: Device: Neuro-muscular electrical stimulation; Procedure: Active exercises
- Functional electrical stimulation (Experimental): Active exercises & Functional electrical stimulation while walking.
  Interventions: Device: Functional electrical stimulation; Procedure: Active exercises

INTERVENTIONS:
Device: Functional electrical stimulation — Electrical stimulation that cause muscle contraction while walking
  Arms: Functional electrical stimulation
Device: Neuro-muscular electrical stimulation — Electrical stimulation that cause muscle contraction in a stationary position
  Arms: Neuro-muscular electrical stimulation
Procedure: Active exercises — Subjects will receive training exercise according to ACL reconstruction protocol

SUMMARY:
The purpose of this study is to examine the short term effect of functional electrical stimulation treatment versus neuro-muscular electrical stimulation on gait quality for patient after anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
Background: Quadriceps weakness is common following anterior cruciate ligament (ACL) reconstruction. The inadequate quadriceps strength contributes to altered gait patterns following ACL reconstruction. Neuromuscular electrical stimulation (NMES) has been shown to reduce quadriceps atrophy post-ACL reconstruction. However, the effect of functional electrical stimulation (FES), a modulation of NMES which enables quadriceps stimulation synchronized with gait, has not been tested.

Objective: The aim of this study is to evaluate the effectiveness of FES to improve the gait pattern of patients post ACL reconstruction.

Methods: Fifty six Individuals post-ACL reconstruction will be randomly placed into FES or NMES treatment group. All patients will receive a standard exercise program three sessions weekly. In addition, each group will receive a different electrical stimulation treatment: Neuromuscular Electrical Stimulation (NMES) or Functional Electrical Stimulation (FES). Outcome measures will include spatiotemporal gait measures (e.g., gait speed, single limb support, and asymmetry index), as well as isometric quadriceps strength. Measures will be taken a week before the surgery, a week after it, and one month from the beginning of rehabilitation. Strength and gait pattern will be measured. Isometric Quadriceps strength will measured using the Biodex isokinetic system, and gait analysis will be carried out through the spatio-temporal Optogait system.

ELIGIBILITY:
* Inclusion Criteria:

  * Intended patients for ACL reconstruction procedure
  * Age 18-30
  * Committed for three sessions per week for 4 weeks
* Exclusion Criteria:

  * Previous surgery at the same knee
  * Chronic knee swelling
  * Knee injury
  * History of recurrent ankle sprains, Achilles tendinopathy, or lower limb

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Percentages of single support at each leg | One year
  The test will perform with the Optogait system (a device for the Gait Analysis). Single support phase within the gait cycle during which the body mass is carried by a single limb. This parameter calculated by percentage of stride (normally about 40%).

SECONDARY OUTCOMES:
strength symmetry | One year
  The method of assessment for this Outcome Measure is by calculated the differences between the right Quadriceps strength and the left Quadriceps strength
Gait speed | One year
  Measured by kilometer per hour
Step length | One year
  Measured by length of the average step for each leg
Quadriceps strength | One year
  Measured by maximal peak torque in each leg (through Biodex Isokinetic dynamometer)

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Springer, Ph.d, Principal Investigator — Physiotherapy department, school of Health Sciences, Ariel University, ISRAEL
Locations (1):
- Zrifin, Rishon LeZiyyon, Doar Tsvai, Israel

IPD SHARING:
Plan to Share IPD: No